CLINICAL TRIAL: NCT01875458
Title: Biomarker Identification in Orthopaedic and Oral Maxillofacial Subjects
Brief Title: Biomarker Identification in Orthopaedic & Oral Maxillofacial Surgery Subjects to Identify Risks of Bisphosphonate Use
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 815570; 815570 (Other: UPenn IRB)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Osteoporosis, With or Without Treatment; Bisphosphonate Treatment; Atypical Femur Fracture; Bisphosphonate Related Osteonecrosis of the Jaws (BRONJ); Healthy Volunteers
Keywords: Aclasta; Actonel; alendronate; alendronate/cholecalciferol; Aredia; Atelvia; Boniva; Didronel; etidronate; Fosamax; Fosamax Plus D; ibandronate; pamidronate; Reclast; risedronate; Skelid; tiludronate; zoledronic acid; Zometa; Bisphosphonate; Atypical Femur Fracture (AFF); Osteoporosis; Bisphosphonate Related Osteonecrosis of the Jaw (BRONJ)
MeSH Terms: conditions — Osteoporosis; Bisphosphonate-Associated Osteonecrosis of the Jaw

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva has been collected from participants and DNA analysis will be performed. Blood and tissue samples has been collected from in-person participants. DNA and RNA analysis will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CASES: Adults with current or past history of bisphosphonate treatment (exposed) with Bisphosphonate related Osteonecrosis of the Jaws (BRONJ), or, Adults with current or past history of bisphosphonate treatment (exposed) with atypical fracture
- COUNTER MATCHED CONTROLS: Adults with current or past history of bisphosphonate treatment (exposed) without bisphosphonate related osteonecrosis of the jaws (BRONJ, or, Adults with current or past history of bisphosphonate treatment (exposed) with typical fracture or joint replacement or osteoporosis
- MATCHED CONTROLS: Adults without current bisphosphonate treatment (unexposed) with Typical fracture (healthy fracture patients) Adults without current bisphosphonate treatment (unexposed) without BRONJ (healthy oral surgery subjects or adults with radionecrosis of the jaws)
- Healthy Adult Volunteers: Healthy volunteers with or without current bisphosphonate treatment without jaw or extremity pathologies or injuries to contribute blood and saliva samples only.

SUMMARY:
Bisphosphonates are drugs that prevent bone loss by blocking the activity of cells that normally resorb bone. The most common examples of these drugs are Boniva and Fosamax. These drugs are available for oral or intravenous dosing and are prescribed at daily, weekly, biweekly, or monthly intervals. Among the many thousands of individuals who currently take these medications, certain individuals experience "atypical" femur fractures preceded by prodromal pain, changes in cortical thickening of bone, or bisphosphonate related osteonecrosis of the jaws (BRONJ). Osteonecrosis of the jaws is defined as exposed bone of the jaws for 8 weeks or more and requires surgical treatment.

This study will attempt to identify genomic and rna biomarkers that may play a role in differential metabolism of bisphosphonates or indicate tendency toward the severe adverse events associated with these drugs.

DETAILED DESCRIPTION:
Collected specimens were subjected to Affymetrix DMET™ Plus Solution analysis. Manuscript is in preparation.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (male or female) age 18 or over meeting any of the following criteria:
* All participants must be able to provide informed consent for themselves.
* History of BP treatment with or without BRONJ and/or Femur fracture (typical or atypical)
* No History of BP treatment with or without BRONJ and/or Femur fracture (typical or atypical)

Exclusion Criteria:

* Children age 17 or younger
* Adults who cannot or do not make medical decisions for themselves
* Persons known to be under the jurisdiction of the Department of Corrections
* Individuals who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who either have ever taken bisphosphonates (see list under Key Words) and/or who have ever had an atypical femur fracture or bisphosphonate related osteonecrosis of the jaws (BRONJ) or both. Also healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2012-04-13 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Absorption, Distribution, Metabolism, Excretion (ADME) Profiling of DNA from all sample types vs. normative data for the ADME panel and across study groups | Baseline
  DNA analysis of saliva, blood, and tissues to detect differential response to drugs. DNA will be isolated from each sample and ADME profiling will be performed. Each participant subgroup will be compared to each other using ANOVA modeling. Each participant subgroup will be compared to normative data for the distribution of gene profiles in the general population for each probe on the ADME gene array.

SECONDARY OUTCOMES:
Differential expression of miRNA biomarkers across participant groups within the study | Baseline
  The relative abundance of miRNA across each participant subgroup will be compared using ANOVA modeling. Each participant subgroup will be compared to normative data for the distribution of miRNA expression profiles in the general population for each probe when available.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Mehta, MD, Principal Investigator — University of Pennsylvania, Department of Orthopaedic Surgery; Annamarie D Horan, PhD, Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
The results of this study will be shared in the form of a published article if accepted. Currently, the manuscript is in draft form and pending submission.